CLINICAL TRIAL: NCT03243201
Title: The Efficacy and Safety of Intranasal Colloidal Silver Nanoparticles for Chronic Rhinosinusitis: A Proof-Of-Concept, Double-Blinded, Placebo-Controlled, Randomized Trial
Brief Title: Silver Nanoparticle Investigation for Treating Chronic Sinusitis
Acronym: SNITCH
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: IND not approved
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 159084
Record Dates: First submitted 2017-08-04; First posted 2017-08-08 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colloidal Silver (Experimental): The colloidal silver arm will administer intranasal colloidal silver, 2 sprays each nostril twice daily, for a total volume of 0.8ml per day (8 mcg of silver per day), for 28 days.
  Interventions: Drug: Colloidal silver nanoparticles
- Purified Water (Placebo Comparator): The placebo arm will administer intranasal purified water, 2 sprays each nostril twice daily, for a total volume of 0.8ml per day, for 28 days.
  Interventions: Other: Purified Water

INTERVENTIONS:
Drug: Colloidal silver nanoparticles — Contains 10ppm colloidal silver nanoparticles
  Other Names: Sovereign Silver, Bio-Active Silver Hydrosol
  Arms: Colloidal Silver
Other: Purified Water — Purified water will be given as placebo
  Arms: Purified Water

SUMMARY:
Chronic rhinosinusitis is a highly prevalent disease resulting in high economic burden. Effective therapeutic options are needed. Rhinosinusitis-related biofilms are a likely contributor to recalcitrant disease. Emerging evidence shows that colloidal silver nanoparticles may be effective for reducing biofilms. The investigators intend to perform a randomized, double-blinded, placebo-controlled clinical trial to evaluate the effectiveness and safety of intranasal colloidal silver nanoparticles in adult patients with chronic rhinosinusitis. The investigators hypothesize that compared to placebo, treatment with intranasal colloidal silver for chronic rhinosinusitis will lead to a significant improvement in symptom scores and will not be associated with increased rate of adverse effects.

ELIGIBILITY:
Inclusion Criteria:

Twelve (12) weeks or longer of two or more of the following signs and symptom consistent with chronic rhinosinusitis (CRS):

* mucopurulent drainage (anterior, posterior, or both), nasal obstruction (congestion), facial pain-pressure-fullness, or decreased sense of smell

AND inflammation is documented by one or more of the following findings:

* purulent (not clear) mucus or edema in the middle meatus or ethmoid region
* polyps in nasal cavity or the middle meatus
* and/or radiographic imaging showing inflammation of the paranasal sinuses

Exclusion Criteria:

* Unable to speak English
* History of nasal or sinus surgery within past 6 weeks
* History of comorbid ciliary dyskinesia, cystic fibrosis or any other mucociliary condition
* Dependence on prolonged corticosteroid therapy for comorbid condition
* History of renal impairment
* History of cerebrospinal fluid leak

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Sino-Nasal Outcome Test (SNOT-22) | Four weeks
  Assess change in SNOT-22 score

IPD SHARING:
Plan to Share IPD: No